CLINICAL TRIAL: NCT00458471
Title: Evaluate the Safety in Human Subjects of Using Bladder Catheters That Are Pre-Coated With a Biofilm That Contains Living Bacteria Escherichia Coli 83972.
Brief Title: E. Coli for Prevention of Catheter UTI in SCI Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Non-Randomized | Purpose: Prevention
Other Study IDs: H-11717
Record Dates: First submitted 2007-04-09; First posted 2007-04-10 (Estimated); Last update posted 2007-04-10 (Estimated); Status verified 2007-04

CONDITIONS: Urinary Tract Infection(UTI)
Keywords: Urinary Catheter; Spinal Cord Injury; Escherichia Coli; Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections; Spinal Cord Injuries; Escherichia coli Infections

INTERVENTIONS:
Device: Insertion of a urinary catheter coated with benign E. coli

SUMMARY:
The overall goal of this project is to develop a new approach for the prevention of urinary tract infection (UTI) in persons who rely on indwelling catheters for bladder drainage. Veterans with spinal cord injury (SCI) frequently require chronic bladder catheterization. Most individuals with SCI have neurogenic bladders, and the resulting urinary stasis and bladder catheterization predispose them to recurrent UTI.1 The presence of a urinary catheter dramatically increases the risk of UTI, not only through contamination of the urinary tract during catheter changes, but also by the presence of a foreign body in the urethra and bladder. Implanted urinary catheters rapidly acquire a complex, three-dimensional biofilm composed of bacteria, their extracellular products, and components deposited from bodily fluids. The pathogenic organisms in a biofilm continually seed the bladder, leading to bacteriuria and/or UTI.2 Bacterial interference, or using benign bacteria to prevent infection with virulent pathogens,3, 4 may offer a solution to the significant problem of recurrent episodes of UTI in persons with indwelling catheters. Since biofilm formation on a wet implanted device such as a urinary catheter is nearly impossible to prevent,5, 6 we propose instead to manipulate the adherent microbial flora. We propose that inserting urinary catheters than have been pre-inoculated with a benign strain of Escherichia coli (83972) will be an efficient means to colonize the neurogenic bladder with this harmless organism. If successful colonization is achieved in this pilot trial, a larger clinical trial will be designed to test the efficacy of this approach to prevent bladder colonization by pathogenic organisms and thus to prevent UTI.

DETAILED DESCRIPTION:
Evaluate urinary catheters that have been pre-inoculated with E. coli 83972 in a prospective clinical trial in SCI patients who require indwelling catheters for bladder drainage:

1. Evaluate in vivo the safety of urinary catheters that have been pre-inoculated with E. coli 83972.
2. Determine whether insertion of such catheters in human subjects can persistently colonize the neurogenic bladder with E. coli 83972. We will define persistent colonization as the presence of E. coli 83972 in the urine for 28 days or longer, as persons with indwelling catheters typically receive a new catheter every 28 days.
3. Evaluate the biofilm present on these urinary catheters after 28 days in the bladder by using both sonication cultures and confocal microscopy.

All patients will have a complete history and physical examination, serum creatinine, plain X-ray of the abdomen, and urine culture immediately prior to entry into the study. Renal ultrasound and urodynamic evaluation of the urinary tract will also be obtained upon study entry unless they have been performed during the preceding year.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed at the Houston VA Medical Center (VAMC) who have sustained spinal cord injury >18 months earlier, suffer from neurogenic bladder, require an indwelling urinary catheter (either transurethral or suprapubic), and do not have vesicoureteral reflux will be enrolled.
* Women and members of minority groups and their subpopulations will be included in this protocol. We anticipate that the gender and minority representation will match the demographic mix for the SCI Unit of the Houston VAMC. We will initially target inpatients for enrollment simply for the patients' convenience, but we will have a low threshold for enrolling suitable outpatients or patients about to be discharged who live close enough to the VAMC to make home visits feasible.

Exclusion Criteria:

* Include urolithiasis, indwelling nephrostomy catheter, supravesical urinary diversion, vesicoureteral reflux, current antibiotic therapy, uncontrolled diabetes mellitus, and immunosuppression.
* Women of childbearing age must have a negative pregnancy test before enrolling in the study, and they must utilize effective birth control methods during the study and for 3 months after the study is concluded.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12
Dates: Start 2003-11; Study Completion 2005-07

PRIMARY OUTCOMES:
bladder colonization and rate of urinary tract infection

CONTACTS AND LOCATIONS:
Overall Officials: Barbara W Trautner, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas, United States

REFERENCES:
- [Result] Stamm WE. Catheter-associated urinary tract infections: epidemiology, pathogenesis, and prevention. Am J Med. 1991 Sep 16;91(3B):65S-71S. doi: 10.1016/0002-9343(91)90345-x. PMID 1928194
- [Result] Costerton JW, Stewart PS, Greenberg EP. Bacterial biofilms: a common cause of persistent infections. Science. 1999 May 21;284(5418):1318-22. doi: 10.1126/science.284.5418.1318. PMID 10334980
- [Result] Sprunt K, Leidy G. The use of bacterial interference to prevent infection. Can J Microbiol. 1988 Mar;34(3):332-8. doi: 10.1139/m88-061. PMID 3046725
- [Result] Stover SL, Lloyd LK, Waites KB, Jackson AB. Urinary tract infection in spinal cord injury. Arch Phys Med Rehabil. 1989 Jan;70(1):47-54. PMID 2644914
- [Result] Habash M, Reid G. Microbial biofilms: their development and significance for medical device-related infections. J Clin Pharmacol. 1999 Sep;39(9):887-98. doi: 10.1177/00912709922008506. PMID 10471979
- [Result] Bastable JR, Peel RN, Birch DM, Richards B. Continuous irrigation of the bladder after prostatectomy: its effect on post-prostatectomy infection. Br J Urol. 1977;49(7):689-93. doi: 10.1111/j.1464-410x.1977.tb04554.x. PMID 597710
- [Result] Thompson RL, Haley CE, Searcy MA, Guenthner SM, Kaiser DL, Groschel DH, Gillenwater JY, Wenzel RP. Catheter-associated bacteriuria. Failure to reduce attack rates using periodic instillations of a disinfectant into urinary drainage systems. JAMA. 1984 Feb 10;251(6):747-51. doi: 10.1001/jama.251.6.747. PMID 6363727